CLINICAL TRIAL: NCT07070115
Title: A Prospective Study Evaluating Clinical Hiatal Hernia Outcomes Using OviTex® Reinforced Tissue Matrix
Brief Title: Evaluating Clinical Hiatal Hernia Outcomes Using OviTex®
Acronym: ECH2O2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tela Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TB_04
Record Dates: First submitted 2025-07-03; First posted 2025-07-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hiatal Hernia
Keywords: hiatal; hernia; reinforced tissue matrix
MeSH Terms: conditions — Hernia, Hiatal; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OviTex Reinforced Tissue Matrix (Other): This is a single-arm study. All study subjects will receive OviTex.
  Interventions: Device: OviTex Reinforced Tissue Matrix

INTERVENTIONS:
Device: OviTex Reinforced Tissue Matrix — All study subjects will receive OviTex. All OviTex Reinforced Tissue Matrices are intended for use as a surgical mesh to reinforce or repair soft tissue where weakness exists.

SUMMARY:
This study will evaluate hiatal hernia recurrence rate and post-operative complications following the use of OviTex Core Resorbable or OviTex 1S Resorbable.

DETAILED DESCRIPTION:
This prospective, open-label, multicenter, non-randomized, post-market study will enroll up to 173 subjects in the United States. Patients undergoing an elective hiatal hernia repair and who meet all eligibility criteria will be enrolled in the study. Subjects will undergo minimally invasive procedures for hiatal hernia repair with the use of OviTex Core Resorbable or OviTex 1S Resorbable for reinforcement. Subjects will have clinical follow-up through 5 years. Data collected in this study will be compared to a literature control at 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a candidate for an elective robotic or laparoscopic primary hiatal hernia repair with the use of OviTex Core Resorbable or OviTex 1S Resorbable.
2. Patient is willing and able to voluntarily sign the IRB-approved Informed Consent Form for the study.
3. Patient is at least 22 years old at the time of surgery.
4. Patient is not pregnant and not planning to become pregnant during the duration of the study (5 years).
5. Patient is able and willing to comply with the study requirements including completion of patient questionnaires and clinic evaluations.

Exclusion Criteria (Baseline):

1. Patient has a Body Mass Index (BMI) of ≥ 35.
2. Patient meets the Centers for Disease Control (CDC) Surgical Site Infection (SSI) Wound Classification Class IV (Dirty-Infected) criteria.
3. Patient has a Type I hiatal hernia (defined as only the esophagogastric junction is above the diaphragm).
4. Patient has a life expectancy of less than five years making it unlikely that the subject will successfully achieve five-year follow-up.
5. Patient is a current nicotine user (including smokeless, vaporized, etc.)
6. Patient has a history of illicit drug or alcohol abuse (in the last three years).
7. Patient has an allergy to ovine-derived products or a known sensitivity to polyglycolic acid (PGA).
8. Patient has an allergy to barium.
9. Patient's surgery will include the use of an anti-reflux implantable device (LINX, etc.).
10. Patient's surgery requires the use of an additional mesh device or a pledget for reinforcement.
11. Patient has participated in another gastrointestinal (GI) clinical study within the past 30 days or is currently involved in another clinical study excluding observational and registry studies.
12. Patient had previous surgery at the gastroesophageal junction.
13. Patient had a prior hiatal hernia repair.
14. Patient has an incarcerated hernia that requires emergent intervention.
15. Patient is a prisoner.

Exclusion Criteria (Intra-operative):

1. Patient is unable to receive OviTex Core Resorbable or OviTex 1S Resorbable at time of surgery.
2. Surgery requires the use of an additional mesh device or a pledget for reinforcement.
3. Surgery includes the use of an anti-reflux implantable device (LINX, etc.).
4. Surgery performed as an open procedure.
5. Patient has a condition, which in the Investigator's opinion, may put the patient at increased risk, confound study data, or interfere significantly with the patient's participation in the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence | At 24 months
  Incidence of radiographic recurrence at 24 months, defined as > 2cm above the hiatus via barium swallow.

SECONDARY OUTCOMES:
Early post-operative complications | Occurring within the first 3 months of the hiatal hernia repair
  Incidence of early post-operative device-related complications noted at the hernia repair site occurring ≤ 90 days after index hiatal hernia repair

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of South Alabama Health, Mobile, Alabama
  - The University of Texas at Austin - Dell Medical School, Austin, Texas

IPD SHARING:
Plan to Share IPD: No